CLINICAL TRIAL: NCT03263104
Title: Single-centre, Prospective, Randomised, Placebo-controlled, Parallel-group Design to Determine the Cholesterol-lowering Efficacy of Lactobacillus Plantarum ECGC 13110402 in Normal to Mildly Hypercholesterolaemic Adults
Brief Title: The Cholesterol-lowering Efficacy of Probiotic Lactobacillus Plantarum in Hypercholesterolaemic Adults
Acronym: PROBIOCHOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, Health Sciences Research Centre, Life Science Department, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UREC 15/06
Record Dates: First submitted 2017-08-17; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Healthy
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Single-centre, prospective, randomised, placebo-controlled, parallel-group design to determine the cholesterol-lowering efficacy of Lactobacillus plantarum ECGC 13110402 in normal to mildly hypercholesterolaemic adults
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind (Participant, Investigator,Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus plantarum ECGC 13110402 (Experimental): Lactobacillus plantarum ECGC 13110402 equivalent to 2x10^9 CFU (0.1 g) with the addition of filling carrier (0.12 g; 30% w/v maltodextrin and 5% w/v sucrose) as a capsular format (vegetable) to be consumed twice daily, before breakfast and dinner with 250mL of water.
  Interventions: Dietary Supplement: Lactobacillus plantarum ECGC 13110402
- Maltodextrin (Placebo Comparator): Maltodextrin (an oligosaccharide without prebiotic effect) (0.12 g; 30% w/v maltodextrin and 5% w/v sucrose) as a capsular format (vegetable) to be consumed twice daily, before breakfast and dinner with 250mL of water.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum ECGC 13110402 — Lactobacillus plantarum ECGC 13110402
  Arms: Lactobacillus plantarum ECGC 13110402
Dietary Supplement: Maltodextrin
  Arms: Maltodextrin

SUMMARY:
Coronary heart disease (CHD) is one of the major causes of death and disability in industrialised countries. Results from several epidemiological and clinical studies indicate a positive correlation between elevated total serum cholesterol levels, mainly reflecting the LDL-cholesterol fraction, and risk of CHD. It is thought that a reduction in total plasma cholesterol levels in populations suffering from primary hypercholesterolemia (elevated cholesterol) can lower the incidence of coronary thrombosis. Currently, therefore there is extensive interest in the management of serum cholesterol and other blood lipids. Diet is viewed as a major influencing factor that can reduce levels. This is largely driven by the expense of drug therapy, the large numbers of individuals affected and unwanted side effects of such treatments. Dietary strategies for prevention of CHD implicate adherence to a low-fat/low-saturated fat diet. Although such diets may present an effective approach, they are difficult to maintain on a long-term basis and efficacy diminishes over time. As such, new approaches towards identification of other dietary means of reducing blood cholesterol levels have been evaluated. These include, among others, the use of probiotics. Probiotics are 'live microbial feed supplements that offer a benefit to health'. They are marketed as health or functional foods whereby they are ingested for their purported positive advantages in the digestive tract and/or systemic areas like the liver, vagina or bloodstream. The main goal of the study was to test whether probiotics can directly degrade cholesterol as well as produce metabolites that interfere with its synthesis in the liver. The effect may also be partially ascribed to an enzymatic deconjugation of bile acids.

DETAILED DESCRIPTION:
The aim of this human volunteer study was to establish tolerance, and the extent of the cholesterol lowering potential of Lactobacillus plantarum ECGC 13110402 in 49, healthy, normal to mildly hypercholesterolaemic adults (30-65 years old).

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 50 years of age.
* in good general health, defined as no comorbidities requiring regular
* medical follow up
* ability to communicate well with the investigator and to comply with the
* requirements of the entire study
* BMI 18.5 to 29.9 kg/m2
* total cholesterol (TC) between 200 and 300 mg/dl (5.16 and 7.64 mmol/L).

Exclusion Criteria:

* History or evidence of organic disease of the gastrointestinal tract; such as tumour, irritable bowel syndrome, etc., within the previous 5 years
* Consumed probiotic or prebiotic preparations on a regular basis (at least 3
* times per week) in the last 2 weeks and during the trial period
* Former participation in another study involving prebiotic or probiotic
* preparations or investigational drugs within the previous 6 months, or
* intention to use such drugs during the course of the study
* high blood cholesterol or use of cholesterol lowering drugs
* Undergone surgical resection of any part of the bowel
* History of malignancy within the previous 5 years (with exception of well-
* treated basal cell carcinoma or in situ cervical carcinoma).
* Currently prescribed immunosuppressive drugs
* Intention to use regularly other medication which affects gastrointestinal
* motility and/or perception
* Current or recent history (within 12 months) of significant drug or alcohol
* abuse or dependence

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Modulation of the blood lipids by L. plantarum ECGC 13110402 The modulation of the blood lipids by L. plantarum ECGC 13110402 | Changes from baseline to 6-12 week treatment period with the probiotic
  Effects of the probiotic on TC, LDL-C, HDL-C and TAG

SECONDARY OUTCOMES:
Modulation of immune function by L. plantarum ECGC 13110402 | Changes from baseline to 6-12 week treatment period with the probiotic
  Blood samples analysis to assess changes in cytokines production Blood samples analysis to assess changes in cytokines production Blood samples analysis to assess changes in cytokines production

OTHER OUTCOMES:
Digestive symptoms | Changes from baseline to 6-12 week treatment period with the probiotic
  Bristol diary form Bristol diary form
Microbiota changes | Changes from baseline to 6-12 week treatment period with the probiotic
  DNA profiling from faeces

CONTACTS AND LOCATIONS:
Overall Officials: Glenn R Gibson, Study Director — The University of Reading

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costabile A, Buttarazzi I, Kolida S, Quercia S, Baldini J, Swann JR, Brigidi P, Gibson GR. An in vivo assessment of the cholesterol-lowering efficacy of Lactobacillus plantarum ECGC 13110402 in normal to mildly hypercholesterolaemic adults. PLoS One. 2017 Dec 11;12(12):e0187964. doi: 10.1371/journal.pone.0187964. eCollection 2017. PMID 29228000